CLINICAL TRIAL: NCT01600027
Title: Effects of Dexmedetomidine Addition to Bupivacaine on the Quality of Fascia Iliaca Compartment Block (FICB) in Children Undergoing Femur Fracture Surgery
Brief Title: Dexmedetomidine Addition to Fascia Iliaca Compartment Block
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Clinical Associate Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R 54; R-54 (Other: Anestheia Dept., Mansoura University)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Children With Fracture Femur
Keywords: Fascia iliaca block; dexmetomidine; fracture femur; α2 agonist
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Placebo Comparator): received 1 ml/kg bupivacaine 0.25%.
  Interventions: Procedure: Fascia iliaca compartment block
- group BD (Active Comparator): received 1 ml/kg bupivacaine 0.25% with dexmedetomidine 2 μg/kg
  Interventions: Procedure: Fascia iliaca block

INTERVENTIONS:
Procedure: Fascia iliaca compartment block — Fascia iliaca compartment block was performed as described by Dalens et al technique.
  Arms: Group B
Procedure: Fascia iliaca block — Fascia iliaca compartment block was performed as described by Dalens et al technique.
  Arms: group BD

SUMMARY:
Fractures of the shaft of femur (FSF) are common in children, especially isolated fractures of the mid-third of the femur which are intensely painful. The pain of the fracture is thought to originate from the femoral shaft periosteum and muscle spasm from the quadriceps mechanism. Fascia iliaca compartment block FIC is easy and simple technique, there is no need for high-skill or expensive equipments. It has higher success rate in more than 90%of the children thigh procedures.

Potentially dexmedetomidine has become an alternative to clonidine, it is a highly selective α2 agonist having about an 8-10 times affinity for α2 adrenergic receptors than clonidine and much less α1 effects, which is responsible for the hypnotic and analgesic effects. Perinural dexmedetomidine in combination with bupivacaine or ropivacaine enhance sensory and motor block without neurotoxicity in experimental studies.It has been reported to improve the quality of intrathecal, Epidural, and caudal anesthesia in children. Also, it is safe and effective in IV regional anesthetic and axillary block in adult. No study-up to the date -has been carried to evaluate its effect on the character of fascia iliaca compartment blocks as adjuvant to bupivacaine. The objectives of this study were designed to detect the effects of addition dexmedetomidine (Precedex- Abbot) as adjuvant to bupivacaine for fascia iliaca block on the quality of postoperative analgesia and also to determine its effects on the hemodynamics, recovery behaviors, sedation and possible side effects in children undergoing thigh surgeries (fracture femur).

DETAILED DESCRIPTION:
All the patients were premedicated with oral midazolam 0.5 mg/kg,1 hour prior to induction. General anesthesia was induced by inhaled sevoflurane.

Laryngeal mask airway with appropriate-size for body weight was slipped, then an intravenous line was inserted,anesthesia was maintained with sevoflurane (Minimum Alveolar Concentration (MAC)from 1-1.5 in air/oxygen to maintain the Heart rate (HR) and mean arterial blood pressure (MAP) within 20% of their baseline values.

A rescue dose of fentanyl 0.5 µg/kg was given if the MAC of sevoflurane exceeded 1.7 whereas HR and MAP exceeded 20% of their baseline values.

Fascia iliaca compartment block was performed as described by Dalens et al technique.

An axillary nerve block needle was inserted with an angle of 45±60º with the skin at (0.5±1cm) below the inguinal crease at the junction of the medial two-thirds and the lateral one-third of the line between the pubic tubercle and anterior superior iliac spine.

The needle was advanced until the perception of two losses of resistance (pop) was noted which corresponded to the crossing of fascia lata and then fascia iliaca.

Hypotension was defined as systolic arterial pressure 70 plus twice the age in years and associated with altered peripheral perfusion.

Bradycardia was defined as HR below 80 beats/min. Delayed anesthetic emergence was defined as 20 min elapsing from the end of surgery to exiting the operating theater.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-6 years
* American Society of Anesthesiologist physical class I and II
* Fracture femur surgery

Exclusion Criteria:

* known allergy to the study drugs
* suspected coagulopathy
* infection at the site of the block
* neurological diseases
* history of developmental delay

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | every 4 hours after surgery
  Postoperative using the Objective Pain Scale (children <6 yr) which described by Hannallah et al.

SECONDARY OUTCOMES:
Vital signs | before surgery, and every 20 min during surgery, and each 6 hours after surgery
  Heart rate, mean arterial pressure and oxygen saturation
Intraoperative hypotension | for 24 hours after surgery
Intraoperative bradycardia | for 24 hours after surgery
Postoperative sedation | every 4 hours after surgery
  Sedation score was assessed using Ramsay's sedation

CONTACTS AND LOCATIONS:
Overall Officials: Ghada F E l-Rahmawy, MD, Principal Investigator — Anesthesia and Surgical ICU, College of Medicine, Mansoura University, Mansoura City, Egypt
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt